CLINICAL TRIAL: NCT03009175
Title: Patient Risk Triage in ICD Remote Follow-up Observational Study (PRoMOTE FU)
Brief Title: PRoMOTE Follow-up Observational Study
Acronym: PRoMOTE FU
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: PRoMOTE FU
Record Dates: First submitted 2016-01-11; First posted 2017-01-04 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantable Cardiac Defibrillator, Cardiac Resynchronization Therapy Defibrillator/Pacemaker

SUMMARY:
The purpose of the study is:

* To evaluate the Heart Failure Risk Status (HFRS) feature performance.
* To establish the feasibility of remote follow-up in which patient risk triaging is performed by nurse-led review of HFRS feature as supplemental information.

ELIGIBILITY:
Inclusion Criteria:

Patients that meet all of following criteria could be included in the study:

* Implant of a commercially available Medtronic CRTD or ICD device with or without the Optivol Fluid Status Monitoring feature.
* Inclusion in the Medtronic Carelink Network.
* Local consent available for CL network as well as general local consent available for the use of data in observational studies signed and informative sheet delivered.

Exclusion Criteria:

* Patients under the age of 18 years.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients of both sexes included in the Medtronic CareLink® Network and implanted with a Medtronic wireless implantable cardiac defibrillator (ICD) or cardiac resynchronization therapy device with defibrillation capabilities device (CRT-D) at Hospital Araba (former Hospital Txagorritxu). There are approximately 223 ICD and CRT-D patients included in the CareLink® Network at this site, and average number of transmissions per month is ~80, so it is expected that 480 transmissions are received during the study duration.
  From this population, less than 10% are implanted with a device without Optivol® feature. For these patients we will not have HFRS data.
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Clinical Data collected through the phone call to the patients during the 6 months of study duration will be correlated to the HF risk classification provided by the HFRS feature on each transmission. | 6 months

IPD SHARING:
Plan to Share IPD: Undecided